CLINICAL TRIAL: NCT04617795
Title: Evaluating the Safety and Effectiveness of the Omnipod® 5 Automated Insulin Delivery System in Patients With Type 2 Diabetes
Brief Title: Omnipod® 5 Automated Insulin Delivery System in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: OP5 in T2D Study G190270
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2D; Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Basal-Bolus (Group A) (Experimental): * 2 weeks standard therapy - using multiple daily injections (MDI) and Dexcom G6 Continuous Glucose Monitor (CGM), followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with optional bolus, followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with simplified bolus
  * 6-month optional extension using Automated Mode
  Interventions: Device: Omnipod 5 Automated Insulin Delivery System
- Basal (Group B) (Experimental): * 2 weeks standard therapy - using basal injection only and Dexcom G6 Continuous Glucose Monitor (CGM), followed by:
  * 2 weeks Omnipod 5 system use in Manual Mode with Dexcom G6 Continuous Glucose Monitor (CGM) - with fixed basal rate, no bolus, followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with optional bolus, followed by:
    * If % time in range 70-180 mg/dL during Automated Mode is ≤50%, 4 weeks Omnipod 5 system use in Automated Mode with simplified bolus, OR
    * If % time in range 70-180 mg/dL during Automated Mode is >50%, 4 weeks Omnipod 5 system use in Automated Mode with optional bolus
  * 6-month optional extension using Automated Mode
  Interventions: Device: Omnipod 5 Automated Insulin Delivery System

INTERVENTIONS:
Device: Omnipod 5 Automated Insulin Delivery System — The Omnipod 5 is a single hormone insulin delivery system intended for the management of diabetes in persons requiring insulin. Continuous subcutaneous insulin infusion may be delivered by user-defined settings (manual mode) or automatically adjusted in response to feedback from a continuous glucose monitor (CGM).
  The Omnipod 5 can automatically increase insulin delivery based on sensor glucose values from the continuous glucose monitor (CGM) and can decrease or suspend delivery of insulin when the glucose value falls below or is predicted to fall below predefined threshold values.
  The Omnipod 5 is designed to assist patients with diabetes in achieving glycemic targets set by their health care providers.

SUMMARY:
The study subjects will be separated into 2 groups, depending on their previous insulin therapy with approximately 50% of subjects from each group, continuous glucose monitoring (CGM) naive.

Group A will complete a 2-week Standard Therapy Phase followed by 8 weeks of Omnipod 5 system use.

Group B will complete a 2-week Standard Therapy Phase followed by 10 weeks of Omnipod 5 system use.

Group A and Group B will have an optional 6-month extension of Omnipod 5 system use

DETAILED DESCRIPTION:
Basal-Bolus - Group A (N=12)

* 2 weeks standard therapy - using multiple daily injections (MDI) and Dexcom G6 continuous glucose monitoring (CGM) , followed by:
* 4 weeks Omnipod 5 system use in Automated Mode with optional bolus, followed by:
* 4 weeks Omnipod 5 system use in Automated Mode with simplified bolus
* 6-month optional extension using Automated Mode

Basal - Group B (N=12)

* 2 weeks standard therapy - using basal injection only and Dexcom G6 continuous glucose monitoring (CGM) , followed by:
* 2 weeks Omnipod 5 system use in Manual Mode with Dexcom G6 continuous glucose monitoring (CGM) - with fixed basal rate, no bolus, followed by:
* 4 weeks Omnipod 5 system use in Automated Mode with optional bolus, followed by:

  * If % time in range 70-180 mg/dL during Automated Mode is ≤50%, 4 weeks Omnipod 5 system use in Automated Mode with simplified bolus, OR
  * If % time in range 70-180 mg/dL during Automated Mode is >50%, 4 weeks Omnipod 5 system use in Automated Mode with optional bolus
* 6-month optional extension using Automated Mode

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 18-75 years
2. Diagnosed with type 2 diabetes on insulin therapy by injection: basal-bolus (12 subjects) or basal only (12 subjects) regimens
3. A1C 8.0-12.0%
4. Has not used an insulin pump within 3 months of screening
5. Willing to use only the following types of insulin during the study: Humalog, Novolog, Admelog or Apidra during the study
6. Maximum insulin dose of 200 units/day
7. Stable doses over the last 4 weeks of other glucose-lowering medications as determined by Investigator
8. Willing to wear the system continuously throughout the study
9. Deemed appropriate for pump therapy per investigator's assessment considering previous history of severe hypoglycemic and hyperglycemic events, and other comorbidities
10. Investigator has confidence that the subject has the cognitive ability and can successfully operate all study devices and can adhere to the protocol
11. Must be willing to use the Dexcom App on the Omnipod 5 PDM as the sole source of Dexcom data (except for the Dexcom Follow App) during Automated Mode
12. Subjects scoring ≥ 4 on the Clarke Questionnaire must agree to have an overnight companion, defined as someone who resides in the same home or building as the study subject and who can be available overnight
13. Able to read and speak English fluently
14. Willing and able to sign the Informed Consent Form (ICF)

Exclusion Criteria:

1. A medical condition, which in the opinion of the investigator, would put the subject at an unacceptable safety risk
2. Planned major surgery during the study
3. History of severe hypoglycemia in the past 6 months
4. History of diabetic ketoacidosis (DKA) in the past 6 months, unrelated to an intercurrent illness, infusion set failure or initial diagnosis
5. Diagnosed with a blood dyscrasia or bleeding disorder
6. Plans to receive blood transfusion over the course of the study
7. Currently diagnosed with anorexia nervosa or bulimia
8. Currently on hemodialysis
9. History of adrenal insufficiency
10. Has taken oral or injectable steroids within the past 8-weeks or plans to take oral or injectable steroids during the study
11. Unable to tolerate adhesive tape or has any unresolved skin condition in sensor or pump placement
12. Plans to use insulin other than U-100 insulin during the Omnipod 5 phase of the study
13. Cardiac disease with functional status New York Heart Association Class III or IV or current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the previous 12-months.
14. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD, or implant)
15. Participation in another clinical study using an investigational drug or device other than the Omnipod 5 in the preceding 30-days or intends to participate during the study period
16. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Carlson, MD, Study Chair — International Diabetes Center at Park Nicollet; Anne Peters, MD, Study Chair — Keck School of Medicine of USC
Locations (4):
- United States (4):
  - University of California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Atlanta Diabetes, Atlanta, Georgia
  - International Diabetes Center, Saint Louis Park, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Basal-Bolus (Group A): * 2 weeks standard therapy - using multiple daily injections (MDI) and Dexcom G6 Continuous Glucose Monitor (CGM), followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with optional bolus, followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with simplified bolus
  * 6-month optional extension using Automated Mode
  Omnipod 5 Automated Insulin Delivery System: The Omnipod 5 is a single hormone insulin delivery system intended for the management of diabetes in persons requiring insulin. Continuous subcutaneous insulin infusion may be delivered by user-defined settings (manual mode) or automatically adjusted in response to feedback from a continuous glucose monitor (CGM).
  The Omnipod 5 can automatically increase insulin delivery based on sensor glucose values from the continuous glucose monitor (CGM) and can decrease or suspend delivery of insulin when the glucose value falls below or is predicted to fall below predefined threshold values.
  The Omnipod 5 is designed to assist patients with diabetes in achieving glycemic targets set by their health care providers.
- Basal (Group B): * 2 weeks standard therapy - using basal injection only and Dexcom G6 Continuous Glucose Monitor (CGM), followed by:
  * 2 weeks Omnipod 5 system use in Manual Mode with Dexcom G6 Continuous Glucose Monitor (CGM) - with fixed basal rate, no bolus, followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with optional bolus, followed by:
    * If % time in range 70-180 mg/dL during Automated Mode is ≤50%, 4 weeks Omnipod 5 system use in Automated Mode with simplified bolus, OR
    * If % time in range 70-180 mg/dL during Automated Mode is >50%, 4 weeks Omnipod 5 system use in Automated Mode with optional bolus
  * 6-month optional extension using Automated Mode
  Omnipod 5 Automated Insulin Delivery System: The Omnipod 5 is a single hormone insulin delivery system intended for the management of diabetes in persons requiring insulin. Continuous subcutaneous insulin infusion may be delivered by user-defined settings (manual mode) or automatically adjusted in response to feedback from a continuous glucose monitor (CGM).
  The Omnipod 5 can automatically increase insulin delivery based on sensor glucose values from the continuous glucose monitor (CGM) and can decrease or suspend delivery of insulin when the glucose value falls below or is predicted to fall below predefined threshold values.
  The Omnipod 5 is designed to assist patients with diabetes in achieving glycemic targets set by their health care providers.
Period: Main Study
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Optional 6-month Extension
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Started | 12 | 12
Completed | 12 | 10
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basal-Bolus (Group A) | Basal (Group B) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.6) | 59.4 (7.5) | 60.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35.19 (4.53) | 31.88 (3.84) | 33.54 (4.44)

OUTCOME MEASURES:

1. Primary Outcome: Hyperglycemia
Description: Overall percentage of time ≥250 mg/dL during standard therapy phase and ALL phases of Automated Mode
Time Frame: 8-10 weeks and after 6-month optional extension
Population: In Group B, only 10 subjects completed the extension study.
Measure: Mean (Standard Deviation); unit: Percent of Time (%)
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percent of Time (%)
  Overall ST | 21.5 (16.8) | 33.3 (23.8)
  Overall AUTO | 9.3 (5.6) | 11.7 (11.3)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 12.4 (11.1) | 6.4 (4.8)

2. Primary Outcome: Hypoglycemia
Description: Overall percentage of time <54 mg/dL during standard therapy phase and all phases of Automated Mode
Time Frame: 8-10 weeks and after 6-month optional extension
Population: In Group B, only 10 subjects completed the extension study.
Measure: Mean (Standard Deviation); unit: Percent of Time (%)
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percent of Time (%)
  Overall ST | 0.19 (0.36) | 0.02 (0.07)
  Overall AUTO | 0.05 (0.09) | 0.01 (0.02)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 0.02 (0.02) | 0.04 (0.05)

3. Secondary Outcome: Percent of Time in Range 70-180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: Automated Mode use (8-10 weeks and after 6-month optional extension) will be compared to the standard therapy phase (2 weeks) overall, separately for Group A and Group B
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: Percent of Time (%)
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percent of Time (%)
  Overall ST | 42.8 (20.4) | 30.5 (17.4)
  Overall AUTO | 60.5 (14.3) | 56.6 (17.7)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 58.1 (15.1) | 65.3 (15.2)

4. Secondary Outcome: Percent of Time > 180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: as for outcome 3
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: Percent of Time (%)
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percent of Time (%)
  Overall ST | 56.3 (20.6) | 69.2 (17.6)
  Overall AUTO | 39.3 (14.3) | 43.3 (17.7)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 41.8 (15.2) | 34.5 (15.1)

5. Secondary Outcome: Percent of Time ≥ 300 mg/dL
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: as for outcome 3
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: Percent of Time (%)
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percent of Time (%)
  Overall ST | 8.8 (9.1) | 16.0 (17.3)
  Overall AUTO | 2.2 (1.8) | 4.3 (5.9)
  Overall Exension: number analyzed (Participants) | 12 | 10
  Overall Exension | 4.5 (5.8) | 1.5 (1.4)

6. Secondary Outcome: Percent of Time < 70 mg/dL
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: as for outcome 3
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: Percent of Time (%)
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percent of Time (%)
  Overall ST | 0.91 (1.54) | 0.26 (0.56)
  Overall AUTO | 0.15 (0.13) | 0.08 (0.13)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 0.11 (0.08) | 0.15 (0.22)

7. Secondary Outcome: Standard Deviation
Description: Glucose metric from study continuous glucose monitoring system-measured glucose variability with the standard deviation
Time Frame: as for outcome 3
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
mg/dL
  Overall ST | 58.3 (17.9) | 61.2 (16.2)
  Overall AUTO | 48.0 (8.5) | 49.6 (14.1)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 52.7 (12.5) | 43.6 (9.2)

8. Secondary Outcome: Coefficient of Variation (of Glucose)
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the coefficient of variation (CV). Calculated by dividing the standard deviation of CGM values by the mean CGM values in the observation period.
Time Frame: as for outcome 3
Population: In Group B, only 10 subjects completed the extension.
Measure: Mean (Standard Deviation); unit: Percent coefficient of variation
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percent coefficient of variation
  Overall ST | 29.2 (6.8) | 27.6 (6.5)
  Overall AUTO | 27.3 (3.8) | 27.0 (5.1)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 29.0 (4.3) | 25.6 (4.5)

9. Secondary Outcome: Mean Glucose
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: as for outcome 3
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
mg/dL
  Overall ST | 199.1 (32.5) | 224.6 (40.9)
  Overall AUTO | 175.5 (16.9) | 181.9 (25.0)
  Overall Extension: number analyzed (Participants) | 12 | 10
  Overall Extension | 180.7 (22.7) | 169.6 (16.8)

10. Secondary Outcome: Total Daily Insulin (Units)
Description: Measure of insulin requirements
Time Frame: as for outcome 3
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
units
  ST | 92.4 (44.0) | 30.6 (21.9)
  AUTO | 63.1 (26.4) | 42.1 (38.4)
  Extension: number analyzed (Participants) | 12 | 10
  Extension | 68.7 (28.5) | 38.7 (33.3)

11. Secondary Outcome: Total Daily Insulin (Units/kg)
Description: Measure of insulin requirements
Time Frame: as for outcome 3
Population: In Group B, only 10 subjects completed the extension.
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
units/kg
  ST | 0.89 (0.32) | 0.33 (0.20)
  AUTO | 0.62 (0.23) | 0.45 (0.40)
  Extension: number analyzed (Participants) | 12 | 10
  Extension | 0.68 (0.28) | 0.40 (0.31)

12. Secondary Outcome: Change in Hemoglobin A1c (HbA1c)
Description: Measures average blood sugar levels over the past 3 months
Time Frame: End of study (8-10 weeks) and during extension (21-23 weeks and 24-26 weeks) compared to baseline (Days 57, 147, and 237 (Group A) or Days 71, 161, and 251 (Group B) compared to Day -30
Population: In Group B, only 10 participants completed the extension.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1C
Arm/Group | Basal-Bolus (Group A) | Basal (Group B)
Number analyzed (Participants) | 12 | 12
Percentage of HbA1C
  Baseline | 9.4 (1.0) | 9.5 (0.8)
  End of Main Study | 8.1 (0.8) | 8.1 (0.6)
  End of Extension: number analyzed (Participants) | 12 | 10
  End of Extension | 8.0 (0.7) | 7.5 (0.6)

ADVERSE EVENTS:
Time Frame: Start of standard therapy (-14d to +1d prior to OP5 start) until the end of the extension [251 days +/- 3 days].
Description: Adverse events listed below were collected from the start of standard therapy until the end of the extension.
Groups:
- Basal-Bolus (Group A): * 2 weeks standard therapy - using multiple daily injections (MDI) and Dexcom G6 Continuous Glucose Monitor (CGM), followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with optional bolus, followed by:
  * 4 weeks Omnipod 5 system use in Automated Mode with simplified bolus
  Omnipod 5 Automated Insulin Delivery System: The Omnipod 5 is a single hormone insulin delivery system intended for the management of diabetes in persons requiring insulin. Continuous subcutaneous insulin infusion may be delivered by user-defined settings (manual mode) or automatically adjusted in response to feedback from a continuous glucose monitor (CGM).
  The Omnipod 5 can automatically increase insulin delivery based on sensor glucose values from the continuous glucose monitor (CGM) and can decrease or suspend delivery of insulin when the glucose value falls below or is predicted to fall below predefined threshold values.
  The Omnipod 5 is designed to assist patients with diabetes in achieving glycemic targets set by their health care providers.
- Basal-Bolus (Group A Extension); Basal (Group B Extension): • 6-month optional extension using Automated Mode
  Omnipod 5 Automated Insulin Delivery System: The Omnipod 5 is a single hormone insulin delivery system intended for the management of diabetes in persons requiring insulin. Continuous subcutaneous insulin infusion may be delivered by user-defined settings (manual mode) or automatically adjusted in response to feedback from a continuous glucose monitor (CGM).
  The Omnipod 5 can automatically increase insulin delivery based on sensor glucose values from the continuous glucose monitor (CGM) and can decrease or suspend delivery of insulin when the glucose value falls below or is predicted to fall below predefined threshold values.
  The Omnipod 5 is designed to assist patients with diabetes in achieving glycemic targets set by their health care providers.
Arm/Group | Basal-Bolus (Group A) | Basal (Group B) | Basal-Bolus (Group A Extension) | Basal (Group B Extension)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 2/12 | 1/10
Other Adverse Events (participants affected / at risk) | 1/12 | 3/12 | 6/12 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal-Bolus (Group A) (N=12) | Basal (Group B) (N=12) | Basal-Bolus (Group A Extension) (N=12) | Basal (Group B Extension) (N=10)
Other (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal-Bolus (Group A) (N=12) | Basal (Group B) (N=12) | Basal-Bolus (Group A Extension) (N=12) | Basal (Group B Extension) (N=10)
Prolonged Hyperglycemia (Endocrine disorders) | 1 (2) | 1 (1) | 4 (9) | 0 (0)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Other (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT04617795/Prot_SAP_002.pdf